CLINICAL TRIAL: NCT00515996
Title: Genetic Abnormalities and Changes of Autonomic Nervous System, Serotonin System, and Neuroendocrine System According to Pharmacotherapy in Panic Disorder
Brief Title: Genetic Abnormalities and Biological Changes of Panic Disorder Patients After Pharmacotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Other Study IDs: C-A6-418-2
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Panic Disorder
Keywords: panic disorder; paroxetine; genetic polymorphism; serotonin
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: paroxetine treatment group vs. normal control group

SUMMARY:
We plan to examine genetic polymorphism of catechol-O-methyltransferase in panic disorder and neurobiological changes of panic disorder patients after 12 weeks of pharmacotherapy with paroxetine. We plan to include 40 panic disorder patients and 40 normal control subjects in this study for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Panic disorder

Exclusion Criteria:

* Other major medical or psychiatric illnesses

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-01; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bum-Hee Yu, M.D. & Ph.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea